CLINICAL TRIAL: NCT01708837
Title: Effect of Depth of Total Intravenous Anesthesia Using Propofol on Postoperative Cognitive Dysfunction : A Multi-Center Study
Brief Title: Effect of Depth of Total Intravenous Anesthesia Using Propofol on Postoperative Cognitive Dysfunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ISSDIPR0003
Record Dates: First submitted 2012-10-07; First posted 2012-10-17 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2012-10

CONDITIONS: Cognition Disorders
Keywords: Postoperative Cognitive Dysfunction; Bispectral index
MeSH Terms: conditions — Cognition Disorders; Postoperative Cognitive Complications | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- deep anesthesia group (Other): Propofol infusion rate is titrated to maintain the target BIS values in 30-45
  Interventions: Drug: Propofol
- light anesthesia group (Other): Propofol infusion rate is titrated to maintain the target BIS values in 45-60
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol infusion rate is titrated to maintain the target BIS values

SUMMARY:
The purpose of this study is to investigate whether the depth of anesthesia with propofol affects the incidence of early postoperative cognitive dysfunction

DETAILED DESCRIPTION:
INTRODUCTION

1.1 Rationale for the study

There is a significant relation between postoperative cognitive dysfunction and increasing age, increasing duration of surgery. But, up to now, the effect of the depth of anesthesia on POCD remains controversial. This study is designed to investigate whether the depth of anesthesia affects the incidence of POCD, we will use propofol for total intravenous anesthesia in elderly patients whose depth of anesthesia was monitored and adjusted by bispectral index (BIS). The early and long-term incidence of POCD will be compared between deep and light-anesthesia groups.

1.2 Background

We hypothesize that depth of anesthesia may exert an influence on the early postoperative cognitive dysfunction. One reason that deep anesthesia might protect cognitive function is the prevention of the stress response to noxious stimulation. The noxious stimulation of surgery can induce stress responses whose severity correlates with the intensity of surgery (major versus minor).Light anesthesia with a serious stress response to noxious stimulation may increase the incidence of POCD. Furthermore, major surgery causing a serious stress response can give rise to a higher incidence of early postoperative cognitive dysfunction than minor. This may also prove our hypothesis on the other hand. The elderly patients who received major surgery had a higher incidence of early POCD than those who received minor surgery. A deleterious stress response can be associated with major surgery or light anesthesia, and it can cause excessive production of corticosteroids that target receptors in the cerebral cortex and subcortical nucleus, eventually resulting in neuron injury. This may explain why the elderly has a higher incidence of early POCD after surgery. However, the effect of the depth of anesthesia on POCD remains controversial. Farag E et al. randomized 74 patients to either a low Bispectral Index (BIS) regimen or a high BIS regimen during the surgical procedure. Preoperatively and 4-6 week after surgery, the patients' cognitive status was assessed with a cognitive test battery consisting of processing speed index, working memory index, and verbal memory index. Processing speed index was higher in the low BIS group versus the high BIS group. But no difference was observed in the other two test battery components. Certainly one of the limitations of their data is that the observed difference in cognitive ability occurred in only one of three assessments. Recently, we have made a randomised, double-blind, controlled study to demonstrate that deeper general anesthesia, as defined by a median BIS of 38, when compared with a median BIS of 58, was associated with a reduced incidence of early POCD(at 1 week postoperationly). This study has been published in J Neurosurg Anesthesiol , Volume 23, Number 1, January 2011. as it was just a small sample(n=40) study without considering incidence of long-term POCD, we hope to obtain more reliable data from a multi-center study to investigate whether the depth of total intravenous anesthesia using propofol affects the early and long-term incidence of POCD.

The bispectral index（BIS）can reflect the depth of anesthesia of propofol combined with opioids. In our study, BIS will still be used to provide a reference for the selection of a suitable depth of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided by legal guardians or patients
* Male or female patients between 50 and 70 years of age.
* ASA physical status I or II patients.
* Education Years of patients are more than 6 years.
* The operation going to be received is the first operation in patient's life (a second operation was a risk factor for early post- operative cognitive dysfunction);
* The operation going to be received is presenting for a moderate surgery, such as pulmonary lobectomy, subtotal gastrectomy, prostatectomy and so on.

Exclusion Criteria:

* The patient has the history of neurologic or mental disease.
* The patient has renal dysfunction, serum creatinine >177 mmol/L.
* The patient has an active liver disease.
* The patient has cardiac dysfunction.
* The patient has pulmonary dysfunction.
* The patient has an endocrine disease.
* The patient has a metabolic disease.
* The patient has a history of surgery.
* The patient is going to receive surgery of thyroid, intracranial procedure, joint replacement, major fracture.
* The patient's education history is shown less than 6 years of school.
* The patient is unable to complete neuropsychologic testing.
* The patient has vision dysfunction.
* The patient has auditory dysfunction.
* The operation going to be received is a laparoscopic surgery.
* The patient is hypersensitive to propofol or any other anesthetic agents.
* Involvement in the planning and conduct of the study
* Participation in another drug trial within 28 days prior enrolment into this study

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-01 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
cognitive function score measured by Wechsler memory scale/ Wechsler intelligence scale manual | Three month
  cognitive function test using Wechsler memory scale/ Wechsler intelligence scale manual were administered the day before and 7 days and 3 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Qulian Guo, PhD, Study Director — Xiangya Hospital, Central South University, Changsha, China
Locations (1):
- XiangYa Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Newman S, Stygall.J: Neuropsychological outcome following cardiac surgery. The Brain and cardiac Surgery 2000: 21-49
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Background] Rasmussen LS, Christiansen M, Rasmussen H, Kristensen PA, Moller JT. Do blood concentrations of neurone specific enolase and S-100 beta protein reflect cognitive dysfunction after abdominal surgery?ISPOCD Group. Br J Anaesth. 2000 Feb;84(2):242-4. doi: 10.1093/oxfordjournals.bja.a013410. PMID 10743460
- [Background] Canet J, Raeder J, Rasmussen LS, Enlund M, Kuipers HM, Hanning CD, Jolles J, Korttila K, Siersma VD, Dodds C, Abildstrom H, Sneyd JR, Vila P, Johnson T, Munoz Corsini L, Silverstein JH, Nielsen IK, Moller JT; ISPOCD2 investigators. Cognitive dysfunction after minor surgery in the elderly. Acta Anaesthesiol Scand. 2003 Nov;47(10):1204-10. doi: 10.1046/j.1399-6576.2003.00238.x. PMID 14616316
- [Background] Johnson T, Monk T, Rasmussen LS, Abildstrom H, Houx P, Korttila K, Kuipers HM, Hanning CD, Siersma VD, Kristensen D, Canet J, Ibanaz MT, Moller JT; ISPOCD2 Investigators. Postoperative cognitive dysfunction in middle-aged patients. Anesthesiology. 2002 Jun;96(6):1351-7. doi: 10.1097/00000542-200206000-00014. PMID 12170047
- [Background] Cai YR, Xue ZG, Zhu B: Risk factors contributing to post- operative cognitive dysfunction in elderly patients. The Journal of Clinical Anesthesiology 2006; 22: 608-610
- [Background] Enlund M, Mentell O, Flenninger A, Horneman G, Ronquist G. Evidence of cerebral dysfunction associated with isoflurane- or propofol based anaesthesia for orthognathic surgery, as assessed by biochemical and neuropsychological methods. Ups J Med Sci. 1998;103(1):43-59. doi: 10.3109/03009739809178944. PMID 9789971
- [Background] Casati A, Fanelli G, Pietropaoli P, Proietti R, Tufano R, Danelli G, Fierro G, De Cosmo G, Servillo G; Collaborative Italian Study Group on Anesthesia in Elderly Patients. Continuous monitoring of cerebral oxygen saturation in elderly patients undergoing major abdominal surgery minimizes brain exposure to potential hypoxia. Anesth Analg. 2005 Sep;101(3):740-747. doi: 10.1213/01.ane.0000166974.96219.cd. PMID 16115985
- [Background] Shim TS, Lee JH, Kim SY, Lim TH, Kim SJ, Kim DS, Kim WD. Cerebral metabolic abnormalities in COPD patients detected by localized proton magnetic resonance spectroscopy. Chest. 2001 Nov;120(5):1506-13. doi: 10.1378/chest.120.5.1506. PMID 11713127
- [Background] Farag E, Chelune GJ, Schubert A, Mascha EJ. Is depth of anesthesia, as assessed by the Bispectral Index, related to postoperative cognitive dysfunction and recovery? Anesth Analg. 2006 Sep;103(3):633-40. doi: 10.1213/01.ane.0000228870.48028.b5. PMID 16931673
- [Result] Newman S, Stygall J, Hirani S, Shaefi S, Maze M. Postoperative cognitive dysfunction after noncardiac surgery: a systematic review. Anesthesiology. 2007 Mar;106(3):572-90. doi: 10.1097/00000542-200703000-00023. PMID 17325517
- [Result] Abildstrom H, Rasmussen LS, Rentowl P, Hanning CD, Rasmussen H, Kristensen PA, Moller JT. Cognitive dysfunction 1-2 years after non-cardiac surgery in the elderly. ISPOCD group. International Study of Post-Operative Cognitive Dysfunction. Acta Anaesthesiol Scand. 2000 Nov;44(10):1246-51. doi: 10.1034/j.1399-6576.2000.441010.x. PMID 11065205
- [Result] Ni D, Shi X, Wu X：Incidence of Postoperative Cognitive Dys- function (POCD) in Aged-patients After General Anesthesia. China Anesthesia and Analgesia 2004; 6: 164-166